CLINICAL TRIAL: NCT06131567
Title: Implantoplasty as Adjunct to Combined Surgical Therapy of Peri-Implantitis: A Randomized Clinical Trial
Brief Title: Implantoplasty as Adjunct to Combined Surgical Therapy of Peri-Implantitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Center of Implantology, Oral and Maxillofacial Surgery, Badajoz, Spain (Other)
Responsible Party: Principal Investigator, Alberto Monje, Head, Center of Implantology, Oral and Maxillofacial Surgery, Badajoz, Spain
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18102021
Record Dates: First submitted 2023-11-09; First posted 2023-11-14 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-01

CONDITIONS: Peri-Implantitis
MeSH Terms: conditions — Peri-Implantitis

STUDY DESIGN:
Intervention Model Description: Randomized clinical trials with paired number of subjects
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Implantoplasty (Experimental): Implantoplasty to all the implant surface
  Interventions: Procedure: Implantoplasty
- Implantoplasty on the supracrestal component (Active Comparator): Implantoplasty only in the supra-crestal component and the infra bony hydrogen peroxide
  Interventions: Procedure: Implantoplasty

INTERVENTIONS:
Procedure: Implantoplasty — Implantoplasty as surface decontamination method

SUMMARY:
Implantoplasty entails polishing of the implant surface during the surgical therapy of peri-implantitis. Given the controversy behind implantoplasty as surface decontamination method in the treatment of peri-implantitis, the goal of this clinical trial is to assess the clinical resolution and radiographic bone gain in peri-implantitis sites treated by means of reconstructive therapy (Inteross® + autogenous bone, Sigmagraft, CA, USA) + implantoplasty in combined defects when compared to the extent of implantoplasty along the exposed implant surface upon the clinical resolution and radiographic bone gain in peri-implantitis sites treated by means of reconstructive therapy (Inteross® + autogenous bone, Sigmagraft, CA, USA).

ELIGIBILITY:
Inclusion criteria

* All patients in age of 18 to 80, non-smokers
* With no presence of systemic disease or medication known to alter bone metabolism, and partial or complete edentulous patients that have no active periodontal disease.
* Peri-implantitis defined according to the EFP/AAP consensus meeting
* Combined defect configuration

Exclusion criteria:

* Pregnancy or lactation
* History of or current smokers
* Uncontrolled medical conditions,
* Cement-retained restoration
* Lacking keratinized mucosa (≤2mm) on the lingual or buccal implant sites.

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Rate of disease resolution | 12 months after surgery
  pocket depth <6mm, no bleeding on probing, no suppuration, no progressive bone loss

CONTACTS AND LOCATIONS:
Locations (1):
- Centro de Implantologia Cirugia Oral y Maxilofacial, Badajoz, Spain

IPD SHARING:
Plan to Share IPD: Undecided